CLINICAL TRIAL: NCT01556048
Title: Pilot Study of Behavioral Activation for Prolonged Grief
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anthony Papa (Other)
Responsible Party: Sponsor-Investigator, Anthony Papa, Assistant Professor, University of Nevada, Las Vegas
Organization: University of Nevada, Las Vegas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SA08/09-07
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Complicated Grief; Prolonged Grief Disorder; Major Depressive Disorder; Posttraumatic Stress Disorder
Keywords: Behavior therapy; Bereavement; Complicated grief; Depression; Posttraumatic Stress Disorder
MeSH Terms: conditions — Prolonged Grief Disorder; Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMMEDIATE START GROUP (Experimental): Randomized to participate in Behavioral Activation for pathological grief starting at Week 1 of entry into the study
  Interventions: Behavioral: Behavioral Activation
- DELAY START GROUP (Placebo Comparator): Randomized to participate in Behavioral Activation for pathological grief starting at Week 12 of entry into the study
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral Activation for Major Depressive Disorder (BA; Martell, Addis, & Jacobson, 2001) is based on behavioral theories of depression, which posit that psychopathology occurs when active, goal-directed behavioral repertoires have been either unreinforced or punished. These aversive consequences tend to reinforce escape and avoidance behavior, such as passively ruminating on unmet needs and/or deprivations, rather than actively engaging the environment. BA employs operant conditioning principles to increase active, goal-directed behavioral strategies and decrease passive or avoidant behavioral strategies to help people engage with and obtain adequate reinforcement from their environment. Use of BA was based research suggesting that disengagement/avoidance is related to prolonged pathology after loss

SUMMARY:
The Institute of Medicine identifies Prolonged Grief (PG) as a critical under-addressed public health problem for which are no empirically supported treatments. The purpose of this application is to pilot-test Behavioral Activation (BA) therapy for PG. BA is a well supported, stand alone intervention for depression and recently applied to posttraumatic stress disorder, which reduces rumination and avoidance behaviors that otherwise thwart access to natural rewarding contingencies and resources. The treatment focuses on promoting stable, active routines, self-care behaviors, enhanced self-efficacy, and reengagement with pleasurable activities and significant social resources. Rumination, disengagement, and low self-efficacy are defining features of PG. Further, in response to loss of intimates, the key factors that differentiate resilient people from those that have difficulties adapting is the maintenance or fast resumption of social and occupational functioning. Thus, the main hypothesis of this study is that BA for PG will result in clinically significant reductions in rumination and functional disengagement. This is a preliminary small-scale pilot assessment of potential efficacy and feasibility of completing a large scale study of BA for PG.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for Prolonged Grief Disorder
* must be 21 years old or older
* if taking psychotropic medication, must have been on a stable dose for three or more months prior to study entry

Exclusion Criteria:

* presence of active suicidal or homicidal ideation
* a history of psychotic symptoms
* current participation in psychosocial treatment focused on grief symptoms
* active substance abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in grief symptoms at weeks 12, 24, and 36 post randomization | Assessments occurring in Weeks 1 (Baseline), 12, 24, and 36 post randomization
  Inventory of Complicated Grief-Revised
Change from Baseline in PTSD symptoms at weeks 12, 24, and 36 post randomization | Assessments occurring in Weeks 1 (Baseline), 12, 24, and 36 post randomization
  PTSD Checklist-Specific
Change from Baseline in symptoms of Major Depressive Disorder at Weeks 12, 24, and 36 post randomization | Assessments occurring in Weeks 1 (Baseline), 12, 24, and 36 post randomization
  Depression Anxiety Stress Scales

SECONDARY OUTCOMES:
Change from Baseline in levels of rumination at Weeks 12, 24, and 36 post randomization | Assessments occurring in Weeks 1 (Baseline), 12, 24, and 36 post randomization
  Ruminative Response Scale
Therapy credibility and client expectancy for improvement after treatment | Assessments occurring post-treatment (12 weeks for immediate start group, 24 weeks for delay start group)
  Credibility/ Expectancy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antony Papa, Ph.D., Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States